CLINICAL TRIAL: NCT05470270
Title: An Open-label, Non-comparative, Multicentre Study to Evaluate the Acceptability of a New Paediatric Formulation of Hydroxycarbamide in Children With Sickle Cell Disease.
Brief Title: Acceptability of a New Paediatric Formulation of Hydroxycarbamide in Children With Sickle Cell Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Theravia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIK-FR-22-1
Record Dates: First submitted 2022-07-19; First posted 2022-07-22 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Sickle Cell Disease
Keywords: hydroxycarbamide; pediatric; acceptability
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- New formulation of hydroxycarbamide (Experimental): Single arm study with a single administration of hydroxycarbamide
  Interventions: Drug: Hydroxycarbamide

INTERVENTIONS:
Drug: Hydroxycarbamide — Single administration of the new dispersible form of hydroxycarbamide at the usual dose in children with sickle cell disease who are already treated with the current form of hydroxycarbamide.

SUMMARY:
This is a prospective, interventional, phase II, open-label, multicentre, national, non-comparative study of a single administration of the new dispersible form of hydroxycarbamide at the usual dose in children with sickle cell disease who are already treated with the current form of hydroxycarbamide (Siklos® 100 mg and/or 1000 mg film-coated tablets).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, signed and dated by both parents or by the legally acceptable representative(s) of the children,
* Child with sickle cell disease, treated with 100 mg and/or 1000 mg Siklos® film-coated tablets at the same daily dose for more than 4 weeks,
* Child aged between 2 and 6 years old,
* Parents capable of communicating with the investigator and understanding the requirements and constraints of the study protocol and willing to comply with the study requirements,
* Children affiliated to a social security plan (including universal health coverage) or beneficiary of a similar insurance plan.

Exclusion Criteria:

* Participation in any other clinical study for any other pharmaceutical product within 4 weeks preceding study inclusion,
* Known hypersensitivity or allergy to the excipients,
* Any surgical or medical condition or any significant illness (of which severe hepatic impairment (Child-Pugh classification C), severe renal impairment, toxic ranges of myelosuppression) that, in the opinion of the investigator, constitutes a risk or a contraindication to the participation of the patient to the study, or that may interfere with the objectives, conduct or evaluation of the study.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Acceptability score | At Day 1 (inclusion visit at study drug administration)
  Acceptability score evaluated by the parent(s) of the child (2-6 years old) and by the child (4-6 years old)

SECONDARY OUTCOMES:
Percentage of children with acceptable acceptability score (neutral to positive scores) | At Day 1 (inclusion visit at study drug administration)
  Neutral to positive scores reported by the parent(s) of the child (2-6 years old), and by the child (4-6 years old)
Distribution of the scores related to the ease of administration | At Day 1 (inclusion visit at study drug administration)
  Score reported by parent(s), based on a 5-point Likert scale,
Distribution of the scores related to the ease of preparation including the ease of constitution of the liquid form and the ease to follow the prescription | At Day 1 (inclusion visit at study drug administration)
  Score reported by the parent(s) based on a 5-point Likert scale,
Score related to the usefulness of the dispersible form, compared with the tablets currently used | At Day 1 (inclusion visit at study drug administration)
  Score reported by the parent(s), based on a 5-point Likert scale
Free comments collected by the investigator | At Day 1 (inclusion visit at study drug administration)
  Questions from child/parent, reactions before/after drug intake
Number of adverse events | At Day 1 (inclusion visit at study drug administration)
  Number of adverse events and percentage of patients reporting at least one adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Bérengère Koel, MD, Principal Investigator — Hopital Universitaire Robert-Debre
Locations (3):
- France (3):
  - InterCommunal Hospital Centre of Creteil, Créteil
  - Necker University Hospital, Paris
  - Robert Debré Hospital, Paris

IPD SHARING:
Plan to Share IPD: No